CLINICAL TRIAL: NCT04213638
Title: Randomized Controlled Trial of Single Microneedle Radiofrequency for Moderate-to-Severe Acne Vulgaris
Brief Title: Trial of Single Microneedle Radiofrequency for Moderate-to-Severe Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1120191113
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group：1 (Experimental): Intervention: Other：Single Microneedle Radiofrequency therapy
  Interventions: Other: Single Microneedle Radiofrequency therapy
- Group：2 (Active Comparator): Intervention: Other：Photodynamic therapy
  Interventions: Other: Photodynamic therapy

INTERVENTIONS:
Other: Single Microneedle Radiofrequency therapy — Subjects are treated with three consecutive sessions of Single Microneedle Radiofrequency therapy at 2-week intervals, with a follow-up visit 12 weeks after the final third treatment. Each treatment session took approximately 30-60 minutes.
  Arms: Group：1
Other: Photodynamic therapy — Subjects are treated with three consecutive sessions of Photodynamic therapy at 2-week intervals, with a follow-up visit 12 weeks after the final third treatment.
  Arms: Group：2

SUMMARY:
The purpose of the study is to testify the efficacy of treating moderate-to-severe acne vulgaris with Single Microneedle Radiofrequency, and provide evidence for the hypothesis that "whether Single Microneedle Radiofrequency therapy could be an alternative to photodynamic therapy for moderate to severe acne vulgaris."

DETAILED DESCRIPTION:
The purpose of the study is to testify whether Single Microneedle Radiofrequency is effective for moderate-to-severe acne vulgaris, through treating moderate-to-severe acne vulgaris patient for 1 month, using photodynamic therapy as controlled group, and try to provide clinical evidence for the hypothesis that "whether Single Microneedle Radiofrequency therapy could be an alternative to photodynamic therapy for moderate to severe acne vulgaris."

ELIGIBILITY:
Inclusion Criteria:

1. Consistent with the diagnostic criteria of moderate-to-severe acne vulgaris (IGA3-4) .
2. Age of a subject is older than 14 and is younger than 45.（including 14 and 45）.
3. Did not take any anti-acne treatment in the last 1 month, and did not take part in any clinical trial.
4. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. systemic acne treatment with oral isotretinoin within 6 months or oral antibiotics in the past 1 month;
2. history of facial procedures like dermabrasion, chemical, or laser peels;
3. history of photosensitive diseases, porphyria, or porphyrin sensitivity.
4. With serious protopathy or disease of cardiovascular, liver, renal, gastrointestinal, hematological systems and so on.
5. Pregnant women or women in lactation.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
The reduction rate of number of acne lesions | 16 weeks
  Measure the reduction rate of number of acne lesions at 16 weeks after treatment compared with a baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Xiang Ya Hospital Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Lynn DD, Umari T, Dunnick CA, Dellavalle RP. The epidemiology of acne vulgaris in late adolescence. Adolesc Health Med Ther. 2016 Jan 19;7:13-25. doi: 10.2147/AHMT.S55832. eCollection 2016. PMID 26955297
- [Background] Xing M, Yan X, Sun X, Wang S, Zhou M, Zhu B, Kuai L, Liu L, Luo Y, Li X, Li B. Fire needle therapy for moderate-severe acne: A PRISMA systematic review and meta-analysis of randomized controlled trials. Complement Ther Med. 2019 Jun;44:253-260. doi: 10.1016/j.ctim.2019.04.009. Epub 2019 Apr 28. PMID 31126563
- [Background] Tang X, Li C, Ge S, Chen Z, Lu L. Efficacy of photodynamic therapy for the treatment of inflammatory acne vulgaris: A systematic review and meta-analysis. J Cosmet Dermatol. 2020 Jan;19(1):10-21. doi: 10.1111/jocd.13197. Epub 2019 Oct 25. PMID 31654468
- [Background] Ahn GR, Kim JM, Park SJ, Li K, Kim BJ. Selective Sebaceous Gland Electrothermolysis Using a Single Microneedle Radiofrequency Device for Acne Patients: A Prospective Randomized Controlled Study. Lasers Surg Med. 2020 Jun;52(5):396-401. doi: 10.1002/lsm.23152. Epub 2019 Sep 10. PMID 31502662